CLINICAL TRIAL: NCT03371420
Title: PET Imaging of Subjects Using 124I-PU-AD: A Pilot Study
Brief Title: PET Imaging of Subjects Using 124I-PU-AD
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Company has ceased operations
Sponsor: Samus Therapeutics, Inc. (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Weill Medical College of Cornell University (Other); Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PU-AD-00-001; NCT02751554 (obsolete NCT alias)
Record Dates: First submitted 2017-11-29; First posted 2017-12-13 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2019-06

CONDITIONS: Lymphoma; Solid Malignancy; Alzheimer Disease; Myeloma
MeSH Terms: conditions — Lymphoma; Alzheimer Disease; Neoplasms, Plasma Cell | interventions — Positron-Emission Tomography; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 124I-PU-AD (Experimental): A single dose of 124I-PU-AD will be administered by intravenous (IV) injection
  Interventions: Drug: PU-AD; Device: PET Scan; Other: Blood Draws

INTERVENTIONS:
Drug: PU-AD
Device: PET Scan
Other: Blood Draws

SUMMARY:
This is a first in-human, open-label pilot (microdose) study of the positron-emitting agent 124I-PU-AD in subjects with specific cancer types (solid malignancy, lymphoma, and/or myeloma) and/or Alzheimer's disease.

DETAILED DESCRIPTION:
This first in-human trial of the positron-emitting agent 124I-PU-AD is an open-label pilot (microdose) study. Up to 10 evaluable subjects who have active disease will be enrolled to evaluate the PK, metabolism, biodistribution, and radiation dosimetry of 124I-PU-AD.

Following a 28-day screening period, eligible subjects will return to the clinic on Day 1. A single dose of 124I-PU-AD will be administered by intravenous (IV) injection to subjects.

After 124I-PU-AD tracer injection, PET scans will be performed at 4 time points. At each time-point, an axial body image is acquired on a state-of-the-art PET-CT scanner. A low-dose CT will be obtained immediately-prior to PET imaging, at each time-point. Serial blood samples will also be obtained at multiple time points.

Subjects will be evaluated to ensure that there are no clinically significant ongoing AEs prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a diagnosis of cancer and/or Alzheimer's Disease, meeting trial eligibility criteria as specified below for either disease:

   Cancer:
   1. Subjects with eligible histologic types of cancer. Eligible histologic types of cancer include solid malignancy, myeloma, and lymphoma.
   2. Cancer histology confirmed by pathology.
   3. Cancerous disease is radiologically-measurable or evaluable as defined by published tumor response criteria (including but not limited to RECIST 1.1).

   Alzheimer's:
   1. Established diagnosis of mild-moderate Alzheimer's disease based upon neurological and neuropsychological evaluation following the National Institute on Aging - Alzheimer's disease Association criteria that recently revisited the NINCDS-ADRDA criteria.
   2. Documentation of diagnosis of mild-moderate Alzheimer's disease, as above, by board-certified neurologist.
2. Subjects who have both cancer and Alzheimer's Disease, subjects are considered eligible if they meet all eligibility requirements for either Alzheimer's Disease or cancer patients, as specified above.

Exclusion Criteria:

1. Subject has unacceptable pre-study organ function during screening defined as:

   1. Bilirubin > 1.5 x institutional upper limit of normal (ULN)
   2. AST/ALT >2.5 x ULN
   3. Albumin < 2 g/dl
   4. GGT > 2.5 x ULN (IF Alkaline phosphatase > 2.5 x ULN)
   5. Creatinine >1.5 x ULN or creatinine clearance < 60 mL/min.
2. Subject has history of acute major illness (i.e., unstable cardiovascular condition.)
3. Subject has concurrent participation in any interventional studies within 30 days of first dose of study drug.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of 124I-PU-AD: area under the curve (AUC) | 1 week
Pharmacokinetic profile of 124I-PU-AD: maximum plasma concentration (Cmax) | 1 week
Pharmacokinetic profile of 124I-PU-AD: trough plasma concentration (Cmin) | 1 week
Pharmacokinetic profile of 124I-PU-AD: plasma half-life (T1/2) | 1 week
Pharmacokinetic profile of 124I-PU-AD: time to maximum plasma concentration (Tmax) | 1 week

SECONDARY OUTCOMES:
Incidence of adverse events | 30 days
  Safety of 124I-PU-AD in subjects as assessed by evaluation of the incidence, nature, and severity of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Morgan, MS, JD, Study Director — Sponsor GmbH
Locations (1):
- Memorial Sloan Kettering, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bolaender A, Zatorska D, He H, Joshi S, Sharma S, Digwal CS, Patel HJ, Sun W, Imber BS, Ochiana SO, Patel MR, Shrestha L, Shah SK, Wang S, Karimov R, Tao H, Patel PD, Martin AR, Yan P, Panchal P, Almodovar J, Corben A, Rimner A, Ginsberg SD, Lyashchenko S, Burnazi E, Ku A, Kalidindi T, Lee SG, Grkovski M, Beattie BJ, Zanzonico P, Lewis JS, Larson S, Rodina A, Pillarsetty N, Tabar V, Dunphy MP, Taldone T, Shimizu F, Chiosis G. Chemical tools for epichaperome-mediated interactome dysfunctions of the central nervous system. Nat Commun. 2021 Aug 3;12(1):4669. doi: 10.1038/s41467-021-24821-2. PMID 34344873